CLINICAL TRIAL: NCT04687488
Title: COVID-19: The Study of Aerosol Generation and Droplet Dispersion and Deposition During Naso-gastric Intubation for Gastrointestinal Motility Investigations
Brief Title: Aerosol and Droplet Dispersion During Gastrointestinal Motility Investigations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S64237
Record Dates: First submitted 2020-12-03; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Aerosol Generation and Droplet Dispersion and Deposition During Naso-gastric Intubation for Gastrointestinal Motility Investigations
MeSH Terms: interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescein (Other): Fluorescein dye and ultraviolet (UV) light are used to assess the aerosol contamination during endonasal investigations. We will dilute medical fluorescein vials (FLUORESCEINE 10% Faure; SERB, 40 Avenue George V, 75008 Paris, France) to a concentration of 1% fluorescein in 10ml of normal saline solution. Next, we swab the nasal cavity with a compress soaked (15 droplets with a pipette) in fluorescein and we apply 5 droplets into the nasal cavity and nasopharynx at the beginning of the investigation.
  After coating the nose with fluorescein, the patient will wear a surgical nose-mouth mask and will be positioned in the bed used for HRiM or MII-pH probe insertion. As the MII-pH probe is removed 24h after placement of the probe, prior to this activity the same fluorescein application method (fluorescein drops and a cotton swab) will be used.
  Interventions: Other: Fluorescein; Other: Particle measurement

INTERVENTIONS:
Other: Fluorescein — For droplet visualization, we will use fluorescein, which has been used for many years in medicine for diagnostic purposes and is safe upon topical administration, as a tracer. There are no local or systemic side effects of topical sodium fluorescein (5). Fluorescein is routinely used in the mouth to stain dental plaque (6). Through the lacrimal duct, the nasal cavity is exposed to fluorescein when it is used for ophthalmological purposes (7). Allergic reactions have been described to intravenous injection, which is not part of our trial. In the setting of head-and-neck and otolaryngological surgeries, coating the mouth with fluorescein has been used to quantify droplet spread, to assess for risk of transmission of COVID-19 (8). Hence, fluorescein can be safely applied to nasal and oropharyngeal cavities. We will use a similar approach, coating the nasal cavity, to study droplet spread from the nose during naso-gastric intubation for motility or reflux testing.
Other: Particle measurement — Quantification of aerosol will be done using a medical particle counter, as used for hospital safety measurements.

SUMMARY:
To obtain more knowledge about the generation of aerosol and droplet dispersion and deposition during naso-gastric intubation for gastrointestinal motility investigations

DETAILED DESCRIPTION:
Health care workers (HCW) at the endoscopy unit are at constant occupational risk for many infectious diseases as they perform daily procedures that are believed to generate aerosol and droplets, which may harvest respiratory pathogens. These daily procedures include for example High Resolution Impedance Manometry (HRiM), 24h multichannel intraluminal impedance-pH monitoring (MII-pH) and endoscopic investigations. It is well-known that these procedures may induce cough, and can generate aerosol and droplets (1). Previous research showed that respiratory pathogens can remain dispersed in aerosol for up to 3 hours and droplets with a viral load remain stable on plastic and stainless steel surfaces (2). Furthermore, it is known that high viral loads may be present in the nasal cavity, nasopharynx and the oropharynx (3). The impact of the occupational risk for HCW at the endoscopy unit was confirmed during the peak of the severe acute respiratory syndrome -coronavirus (SARS-CoV) outbreak, as confirmed in an online survey from 39 motility centers in Europe. This survey showed that 35 out of 39 centers reduced their capacity during the SARS-CoV outbreak in the month of March 2020 with a median of 100% (range 50-100%) for esophageal HRiM and with a median of 100% (range 80-100%) for MII-pH (4).

Therefore, with resumption of clinical activities during the recovery phase of the SARS-CoV outbreak, a number of guidelines and measures are taken to protect patients and personnel from viral spread. Patients are screened for SARS-CoV infection by reverse transcription polymerase chain reaction ((RT-)PCR) testing on a nasopharyngeal swab specimen prior to invasive investigations and they are required to wear a chirurgical facemask in the hospital at all times. Staff of the endoscopy and function testing units are wearing a chirurgical facemask, standard gloves, goggles, hairnet and a water-resistant gown. Moreover, patients are required to keep a surgical mask over their mouth during the naso-gastric probe positioning, and the bed is lowered so that the head of the patient is below the neck level of the technician. Throughout the procedure, the technician positions him- or herself to the side and back of the patient. However, there is a lack of scientific evidence on the amount of aerosol and droplet spread when these procedures are being performed, with the safety measures that are outlined (1, 4).

ELIGIBILITY:
Inclusion Criteria:

Aged >18 years old;

* Male or female patients;
* Patients undergoing elective gastrointestinal motility investigations (MII-pH and HRiM);
* Negative PCR on nasopharyngeal swab 24 hours prior to the test;
* No anatomical deformity of nose and throat, no known diseases of nose and throat;
* Signed informed consent.

Exclusion Criteria:

* Females who are pregnant or lactating;
* Use of anticoagulant medication;
* Known allergy to fluorescein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Number of droplets spread on the investigator and their location on gown or goggles, by the end of the procedure of naso-gastric intubation for gastrointestinal motility investigations. | After the motility investigation (within 1 hour)
  Visualization of the number of droplets using a UV-lamp (wood lamp) to detect the spread of droplets.

SECONDARY OUTCOMES:
Generation of aerosol particles by insertion and by removal of the naso-gastric motility or pH monitoring probe. | Before placement of the probe (1 and 5 minutes) and after the removement of the probe (1 and 5 minutes).
  Measurement of the aerosol particles in the room during motility investigations.

CONTACTS AND LOCATIONS:
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided